CLINICAL TRIAL: NCT02527551
Title: Efficacy of Deep Haptic Massage in Fibromyalgia : Preliminary Study
Acronym: FEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-AOI-06
Record Dates: First submitted 2015-07-16; First posted 2015-08-19 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Haptic massage (Other): 6 weeks of deep haptic massage at 2 sessions of 30 minutes per week.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — 6 weeks of deep haptic massage at 2 sessions of 30 minutes per week.

SUMMARY:
Fibromyalgia syndrome (FMS) is a common chronic musculoskeletal pain disorder of unknown etiology, characterized by generalized body pain, hyperalgesia and other functional and emotional comorbidities. Women are predominantly affected. Long term prognosis of FMS might be severe by its physical and psychological consequences. The etiology of FMS remains unknown but recent studies suggest a disorder of central pain modulation, neurotransmitters, sympatho-adrenal and hypothalamic-pituitary-adrenal system and peripheral muscles issues. Indeed, muscular abnormalities with a decrease of ATP and micro vascularization have been reported, inducing muscle weakness and local biochemical changes that participate to pain hyper sensitivity. Treatment of FMS is only symptomatic, often difficult, associating pharmacological and non-pharmacological therapies. Massages are largely used in FMS and are included in chronic pain management recommendations.

Massages are recognized as haptic when the hands of the practitioner move on the skin of the patient; haptic massage is superficial if the pressure applied on the skin is similar to the weight of the hand and it's a deep haptic massage when the pressure applied is over the weight of the hand, allowing reaching deep muscle structure. Deep haptic massages are largely used for athlete to improve muscle recovery and treat tendinitis. All massages evaluate in FMS are superficial haptic massage; they are recognized as efficient on pain, anxiety and depression if they are performed at least on 5 weeks but these effects are transient et remain to be optimized. The efficacy of deep haptic massage has not been evaluated in pathological conditions. The investigators hypothesize that, in FMS patients, deep intramuscular maneuvers may solicit sensitive receptors, stimulating large caliber fibers A lemniscal conveyed by the way that bypass chronic pain information carried by the C fibers of the extra-lemniscal pathway: this is the "Gate Control" theory for inhibiting pain information.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 65 years
* Fibromyalgia defined according to ACR criteria
* Widespread pain index (WPI) ≥ 7 and Symptom Severity (SS) scale score ≥ 5 or WPI between 3 and 6 and SS scale score ≥ 9;
* Presence of symptoms at the same intensity for at least 3 months;
* Available to participate in the proposed sessions six weeks
* Drug Therapy Stable fibromyalgia for one month without amendment in the next 6 months, excluding analgesics
* Having signed an informed consent
* Affiliated to a health insurance plan

Exclusion criteria

* Vulnerable people: pregnant women, and breastfeeding women (a urine pregnancy test will be performed), minors, adults under guardianship, deprived of freedom, those hospitalized without consent, hospitalized in a health and social facility for other purposes as research, people unable to consent
* Chronic Inflammatory joint disease associated
* Other non-pharmacological treatments (acupuncture, cognitive-behavioral therapy etc ...)
* Impairments severe visceral: heart, kidney, liver in the previous year
* Individualized psychiatric pathology
* Current Infectious diseases
* Skin lesions contra-indicating massage

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness measured by QIF (Questionnary Impact Fibromyalgia) score | At the end of 6 weeks of deep haptic massage at 2 sessions of 30 minutes per week.
  To evaluate the effectiveness of the Massage Haptic in 20 women with FMS (defined according to the criteria of the American College of Rheumatology and active disease defined by a Widespread Pain Index (WPI)vscore ≥ 7 and a symptom severity score (SS) ≥ 5 or WPI between 3 and 6 and SS score ≥ 9), recruited in the clinics of the Rheumatology Department of Nice, after 6 weeks of deep haptic massage at 2 sessions of 30 minutes per week.
  Primary endpoint: overall score of impact questionnaire fibromyalgia (QIF). Indeed, in the fibromyalgia studies QIF is used as a criterion for evaluating the effectiveness of drug treatments like non-drug treatments.

SECONDARY OUTCOMES:
Effectiveness on pain measured by items 4 to 10 of QIF score | 3 and 6 months
  To assess the continuing effects at 3 and 6 months and the impact on pain The effectiveness of haptic massage will be evaluated in the same manner as the main objective.
  The effectiveness of haptic massage on pain will be evaluated through the individual analysis of the items 4 to 10 of QIF score. These items are listed by EVA.
Effectiveness on fatigue measured by items 4 to 10 of QIF score | 3 and 6 months
  To assess the continuing effects at 3 and 6 months and the impact on fatigue The effectiveness of haptic massage will be evaluated in the same manner as the main objective.
  The effectiveness of haptic massage on fatigue will be evaluated through the individual analysis of the items 4 to 10 of QIF score. These items are listed by EVA.
Effectiveness on anxiety measured by items 4 to 10 of QIF score | 3 and 6 months
  To assess the continuing effects at 3 and 6 months and the impact on anxiety The effectiveness of haptic massage will be evaluated in the same manner as the main objective.
  The effectiveness of haptic massage on anxiety will be evaluated through the individual analysis of the items 4 to 10 of QIF score. These items are listed by EVA.
Effectiveness on stiffness measured by items 4 to 10 of QIF score | 3 and 6 months
  To assess the continuing effects at 3 and 6 months and the impact on stiffness The effectiveness of haptic massage will be evaluated in the same manner as the main objective.
  The effectiveness of haptic massage on stiffness will be evaluated through the individual analysis of the items 4 to 10 of QIF score. These items are listed by EVA.
Effectiveness on depression measured by items 4 to 10 of QIF score | 3 and 6 months
  To assess the continuing effects at 3 and 6 months and the impact on depression The effectiveness of haptic massage will be evaluated in the same manner as the main objective.
  The effectiveness of haptic massage on depression will be evaluated through the individual analysis of the items 4 to 10 of QIF score. These items are listed by EVA.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane SWEERTVAEGHER, Director, Study Director — CHU of the Nice
Locations (1):
- BREUIL, Nice, France

IPD SHARING:
Plan to Share IPD: No